CLINICAL TRIAL: NCT03713944
Title: A Phase II Study of Carboplatin Plus Pemetrexed Plus Atezolizumab Plus Bevacizumab in Chemotherapy and Immunotherapy-naïve Patients With Stage IV Non-squamous Non-small Cell Lung Cancer: Big Ten Cancer Research Consortium BTCRC-LUN17-139
Brief Title: Carboplatin Plus Pemetrexed Plus Atezolizumab Plus Bevacizumab in Chemotherapy and Immunotherapy-naïve Patients With Stage IV Non-squamous Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Extreme toxicity, thromboembolic events
Sponsor: Nasser Hanna (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Nasser Hanna, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC-LUN17-139
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: NSCLC Stage IV; NSCLC, Recurrent
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Recurrence | interventions — Carboplatin; Pemetrexed; atezolizumab; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Single Arm Therapeutic study using historical controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Carboplatin, Pemetrexed, Atezolizumab plus Bevacizumab (Experimental): Carboplatin (AUC 5) i.v. day 1 plus pemetrexed (500 mg/m2) i.v. day 1 plus atezolizumab 1200 mg i.v. day 1 plus bevacizumab 15 mg/kg i.v. day 1 every 3 weeks for up to 4 cycles.
  Patients with non-PD after 4 cycles will be permitted to continue with maintenance therapy with pemetrexed plus atezolizumab plus bevacizumab every 3 weeks until the time of disease progression or intolerable toxicities.
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin, AUC 5
Drug: Pemetrexed — Pemetrexed 500mg/m2
Drug: Atezolizumab — Atezolizumab 1200mg
Drug: Bevacizumab — Bevacizumab 15mg/kg

SUMMARY:
This is a multicenter single arm phase II clinical trial. All eligible patients will receive:

Carboplatin (AUC 5) i.v. day 1 plus pemetrexed (500 mg/m2) i.v. day 1 plus atezolizumab 1200 mg i.v. day 1 plus bevacizumab 15 mg/kg i.v. day 1 every 3 weeks for up to 4 cycles.

Patients with non-PD after 4 cycles will be permitted to continue with maintenance therapy with pemetrexed plus atezolizumab plus bevacizumab every 3 weeks until the time of disease progression or intolerable toxicities.

DETAILED DESCRIPTION:
The hypothesis of this study is that the addition of Atezolizumab (an anti-PD-L1 antibody), to the combination of Carboplatin plus Pemetrexed plus Bevacizumab, a vascular endothelial growth factor (VEGF) inhibitor, for the treatment of patients with stage IV non-squamous, non-small cell lung cancer (NSCLC) will improve progression free survival (PFS) compared with a historical control of carboplatin plus pemetrexed plus bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 within 28 days prior to registration.
* Must have life expectancy of > 3 months at time of consent
* Histological or cytological confirmation of non-squamous NSCLC.
* Must have known PD-L1 status using the Dako 22C3 antibody (+ vs. -) OR must have at least 5 unstained slides to perform PD-L1 testing (results not required for eligibility). PD-L1 positive is defined as a tumor proportion score (TPS) ≥ 1%. PD-L1 negative is defined as a TPS <1%.
* Patients with known targetable mutations in EGFR or BRAF or known translocations in ALK or ROS1 are eligible if they have received FDA approved targeted therapy first. A 1-week washout prior to enrollment is strongly encouraged (3 weeks preferred).
* Stage IV disease or recurrent disease
* Measurable disease according to RECIST v1.1 criteria within 28 days prior to registration with either PET/CT scan, CT scan of chest and abdomen, or CT chest including upper abdomen and adrenal glands which define stage IV disease.
* Patients who had disease progression greater than 1 year after completing prior adjuvant therapy for stage I - III are eligible as long as no systemic therapy was given for recurrence.
* No prior immunotherapy or antiangiogenic therapy.
* Prior platinum therapy or pemetrexed are permissible if previously given in the adjuvant setting for stage I-III disease and disease recurrence is > 1 year from completion of therapy.
* If subject received major surgery or radiation therapy of > 30 Gy, they must have recovered from the toxicity and/or complications from the intervention.
* Demonstrate adequate organ function as defined below, with all screening labs to be obtained within 28 days prior to registration

  * Absolute Neutrophil Count (ANC) ≥ 1.5 K/mm3
  * Hemoglobin (Hgb) ≥ 9 g/dL
  * Platelets ≥ 100 K/mm3
  * Serum creatinine: ≤1.5 X upper limit of normal (ULN) OR Calculated Creatinine Clearance: ≥ 40 cc/min using the Cockcroft-Gault formula
  * Bilirubin ≤ 1.5 × upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) ≤ 1.5 × ULN or < 5x ULN if the transferase elevation was due to liver metastases
  * Alanine aminotransferase (ALT) ≤ 1.5 × ULN or <5x ULN if the transferase elevation was due to liver metastases
  * International Normalized Ratio (INR) or Prothrombin Time (PT) & aPTT ≤ 1.5 × ULN (unless subjects is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants)
* Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to registration. NOTE: A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (> 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus).
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use two non-hormonal methods of contraception, including at least one method with a failure rate of < 1% per year, during the treatment period and for 5 months after the last dose of atezolizumab or 120 days after the last dose of any study drug, whichever is later;

  * examples of non-hormonal contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. Must use "estrogen-free" hormonal method if this is chosen contraception method.
  * A barrier method may be used as the second contraceptive method. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* Contraception method must begin starting from the time of informed consent until 120 days after treatment discontinuation.
* For men: Agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:
* With female partners of childbearing potential or pregnant female partners, men must remain abstinent or use a condom during the treatment period and for 120 days after the last dose of study treatment to avoid exposing the embryo. Men must refrain from donating sperm during this same period.
* The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study

Exclusion Criteria:

* Active infection requiring systemic therapy
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Active secondary cancers.
* Symptomatic, untreated, or actively progressing central nervous system (CNS) metastases. Brain imaging with either MRI or CT with contrast must be performed on all subjects at screening to evaluate for the presence of brain metastases. Patients with a history of treated CNS lesions are eligible, provided that all of the following criteria are met:

  * Measurable disease, per RECIST v1.1, must be present outside the CNS.
  * The patient has no history of intracranial hemorrhage or spinal cord hemorrhage.
  * Metastases are limited to the cerebellum or the supratentorial region (i.e., no metastases to the midbrain, pons, medulla, or spinal cord).
  * The patient has not received stereotactic radiotherapy within 14 days prior to initiation of study treatment or whole-brain radiotherapy within 21 days prior to initiation of study treatment
  * The patient has no ongoing requirement for corticosteroids as therapy for CNS disease and off steroid therapy for at least 14 days. Anticonvulsant therapy at a stable dose is permitted.
  * Asymptomatic patients with CNS metastases newly detected at screening are eligible for the study after receiving radiotherapy or surgery, with no need to repeat the screening brain scan.
* Major surgery within 3 weeks of the first dose of trial treatment.
* Completed palliative radiotherapy within 7 days of the first dose of trial treatment.
* The patient had a history of uncontrolled hereditary or acquired thrombotic disorder.
* Patients with a history of gross hemoptysis (defined as bright red blood or ≥1/2 teaspoon) within 2 months prior to enrollment.
* The patient had clinically relevant congestive heart failure (CHF; NYHA II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
* The patient had experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to enrollment.
* The patient had uncontrolled arterial hypertension ≥150 / ≥90 mm Hg despite standard medical management.
* The patient has had a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to enrollment.
* Patients with ≥ 2 + protein on dipstick urinalysis. All patients with ≥ 2 + protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection and must demonstrate ≤ 1 g of protein in 24 hours to be eligible.
* Clear cavitation of pulmonary lesions seen on imaging.
* The patient had significant bleeding disorders, vasculitis, or experienced Grade 3-4 gastrointestinal (GI) bleeding within 3 months prior to enrollment.
* History of GI perforation and/or fistulae within 6 months prior to enrollment.
* Evidence of tumor invading or abutting major blood vessels.
* The patient had a bowel obstruction, history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
* Has received a live-virus vaccination within 30 days of planned treatment start. Seasonal flu vaccines that do not contain live virus are permitted.
* Previously had a severe hypersensitivity reaction to treatment with another monoclonal antibody (mAb).
* Has active autoimmune disease that has required systemic treatments in the past 2 years, including but not limited to cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents; chronic or occasional use of low-dose steroid therapy can be still be considered eligible as long as no greater than the daily equivalent of 5mg oral prednisone.
* Exceptions to excluding patients with active autoimmune disease include the following:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations are eligible for the study provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months
* Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study. Subjects on chronic systemic steroids would be excluded from the study.
* Had prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or five half-lives of the drug (whichever is longer) prior to initiation of study treatment
* Treatment with systemic immunosuppressive medication (including, but not limited to corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the course of the study, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
* Treatment with denosumab (a RANKL inhibitor) within 4 weeks prior to initiation of study treatment. Patients receiving denosumab prior to enrollment must be willing and eligible to receive a bisphosphonate during atezolizumab treatment.
* History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Has known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Has known active Hepatitis B or C. Active Hepatitis B is defined as a known positive HBsAg result. Active Hepatitis C is defined by a known positive Hep C Ab result and known quantitative HCV RNA results greater than the lower limits of detection of the assay. For patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBcAb] and absence of HBsAg), the patient is only eligible if they are negative for HBV DNA.
* Active tuberculosis
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Has known interstitial lung disease or history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted. Lymphangitic spread of the NSCLC is not exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasser Hanna, MD, Principal Investigator — Indiana University School of Medicine
Locations (7):
- United States (7):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Indiana Univeristy Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab: Carboplatin (AUC 5) i.v. day 1 plus pemetrexed (500 mg/m2) i.v. day 1 plus atezolizumab 1200 mg i.v. day 1 plus bevacizumab 15 mg/kg i.v. day 1 every 3 weeks for up to 4 cycles.
  Patients with non-PD after 4 cycles will be permitted to continue with maintenance therapy with pemetrexed plus atezolizumab plus bevacizumab every 3 weeks until the time of disease progression or intolerable toxicities.
  Carboplatin: Carboplatin, AUC 5
  Pemetrexed: Pemetrexed 500mg/m2
  Atezolizumab: Atezolizumab 1200mg
  Bevacizumab: Bevacizumab 15mg/kg
Period: Study Treatment
Arm/Group | Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab
Started | 30
Completed | 0
Not Completed | 30
Not completed — Patient non-compliance | 1
Not completed — Alternative Cancer Therapy | 3
Not completed — Disease Progression | 18
Not completed — AE/Side Effects/Complications | 2
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Subject decided to come off study due to hip replacement | 1
Not completed — Symptomatic Deterioration | 2
Period: Follow up
Arm/Group | Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab
Started (Treatment and Follow up both are at different time period. Therefore, the number of subjects to start follow up is not equal to the number of subjects who have completed treatment.) | 30
Completed | 14
Not Completed | 16
Not completed — Withdrawal by Subject | 2
Not completed — Death | 11
Not completed — Study Terminated | 3

BASELINE CHARACTERISTICS:
Arm/Group | Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 64 [38 to 83]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 20
  Gender: Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  RACE: Asian | 3
  RACE: Black or African American | 5
  RACE: Multiple (White and Asian) | 1
  RACE: Unknown | 1
  RACE: White | 20
Disease Status at Study Entry [Count of Participants; unit: Participants] — Stage IV: This stage means that the cancer has spread to other organs or parts of the body. It may be also called advanced or metastatic cancer.
  Recurrent Disease: Recurrent Disease is cancer that returns after a period of complete remission. The same type of cancer cells originally found and treated come back in the same or a different location in the body after at least one year of having no detectable evidence of disease.
  Participants
    Recurrent Disease | 3
    Stage IV | 27
PD-L1 Expression Category(Dako 22C3) [Count of Participants; unit: Participants] — The PD-L1 expression was determined by the Tumor Proportion Score (TPS), the percentage of viable tumor cells showing partial or complete membrane staining at any intensity and classified into TPS <1%: No PD-L1 expression TPS 1 to 49%: Low PD-L1 expression TPS ≥50% : High PD-L1 expression
  Participants
    <1 % | 8
    1-49 % | 15
    >=50 % | 7
Primary Histology [Count of Participants; unit: Participants] — NSCLSC : non- small cell lung cancer NOS : not otherwise specified
  Participants
    Adenocarcinoma | 26
    NSCLC, NOS | 4
Smoking Status [Count of Participants; unit: Participants]
  Former (not actively smoking) | 22
  Never (Less than 100 cigarettes in a lifetime) | 8
Received chemotherapy previously [Count of Participants; unit: Participants]
  No | 24
  Yes | 6
Baseline ECOG [Count of Participants; unit: Participants] — ECOG Performance Status can be described as :
  0 Fully active; no performance restrictions.
  1. Strenuous physical activity restricted; fully ambulatory and able to carry out light work.
  2. Capable of all self-care but unable to carry out any work activities. Up and about >50% of waking hours.
  3. Capable of only limited self-care; confined to bed or chair >50% of waking hours.
  4. Completely disabled; cannot carry out any self-care; totally confined to bed or chair.
  Participants
    0 | 10
    1 | 20
EGFR Mutation testing done [Count of Participants; unit: Participants]
  No | 2
  Yes | 28
ALK Mutation testing done [Count of Participants; unit: Participants]
  No | 4
  Yes | 26
ROS-1 Rearrangement testing done [Count of Participants; unit: Participants]
  No | 7
  Yes | 23
HER-2 Mutation testing done [Count of Participants; unit: Participants]
  No | 23
  Yes | 7
RET Translocation testing done [Count of Participants; unit: Participants]
  No | 12
  Yes | 18
MET Mutation testing done [Count of Participants; unit: Participants]
  No | 12
  Yes | 18
KRAS Mutation testing done [Count of Participants; unit: Participants]
  No | 9
  Yes | 21
NTRK Fusion testing done [Count of Participants; unit: Participants]
  No | 16
  Yes | 14
BRAF Mutation testing done [Count of Participants; unit: Participants]
  No | 5
  Yes | 25
Tumor Mutational Burden [Count of Participants; unit: Participants]
  No | 23
  Yes | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) defined as the time from the initiation of treatment to the time when the criteria for disease progression is met as defined by RECIST v1.1 or death of any cause.Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From C1D1 until progression or death up to maximum of 20 Months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Arm A: Carboplatin (AUC 5) i.v. day 1 plus pemetrexed (500 mg/m2) i.v. day 1 plus atezolizumab 1200 mg i.v. day 1 plus bevacizumab 15 mg/kg i.v. day 1 every 3 weeks for up to 4 cycles.
  Patients with non-PD after 4 cycles will be permitted to continue with maintenance therapy with pemetrexed plus atezolizumab plus bevacizumab every 3 weeks until the time of disease progression or intolerable toxicities.
  Carboplatin: Carboplatin, AUC 5
  Pemetrexed: Pemetrexed 500mg/m2
  Atezolizumab: Atezolizumab 1200mg
  Bevacizumab: Bevacizumab 15mg/kg
Arm/Group | Arm A
Number analyzed (Participants) | 30
months | 11.3 [5.5 to 14.9]

2. Secondary Outcome: Overall Response Rate
Description: Overall Response rate will include confirmed complete response (CR) + confirmed partial response (PR), as determined as per RECIST v1.1 criteria and assessed by the local investigator or designee.
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: From C1D1 until death or up to a maximum of 28 months.
Population: Two patients died prior to first post-baseline assessments.Therefore, 28 out of 30 subjects are analyzed for this objective.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A
Number analyzed (Participants) | 28
percentage of participants | 42.9 [24.5 to 62.8]

3. Secondary Outcome: Disease Control Rate
Description: Disease control rate will include complete response (CR], partial response (PR), and stable disease (SD), as per RECIST v1.1 criteria.
Time Frame: From C1D1 until death or up to a maximum of 28 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A
Number analyzed (Participants) | 28
percentage of participants | 92.9 [76.5 to 99.1]

4. Secondary Outcome: Overall Survival
Description: To estimate the overall survival (OS) of carboplatin plus pemetrexed plus atezolizumab plus bevacizumab in immunotherapy and chemotherapy-naïve patients with stage IV non-squamous non-small cell lung cancer.
Time Frame: From C1D1 up to a maximum of 28 Months or until death
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A
Number analyzed (Participants) | 30
months | 22.4 [15.7 to NA] — Upper limit has not been reached.

5. Secondary Outcome: Number of Participants With Adverse Events
Description: To characterize the toxicity of carboplatin plus pemetrexed plus atezolizumab plus bevacizumab in immunotherapy and chemotherapy-naïve patients with stage IV non-squamous non-small cell lung cancer as defined by the NCI Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.
Time Frame: From C1D1 up to a maximum of 20 Months or until death
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A
Number analyzed (Participants) | 30
Participants
  Patient had at least one adverse event of any grade | 30
  Patient had at least one grade 3 or greater adverse event | 24
  Patient had at least one grade 3 or greater treatment related adverse event | 19
  Patient had serious adverse event | 12

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed from C1D1 up to a maximum of 28 Months or until death. All-Cause Mortality was assessed from C1D1 up to a maximum of 28 Months or until death.
Description: An Adverse Event is any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Arm/Group | Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab
All-Cause Mortality (participants affected / at risk) | 11/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab (N=30)
ANEMIA (Blood and lymphatic system disorders) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 2 (3)
COLONIC PERFORATION (Gastrointestinal disorders) | 1 (2)
CONFUSION (Psychiatric disorders) | 1 (1)
DEATH NOS (General disorders) | 1 (1)
ESOPHAGEAL STENOSIS (Gastrointestinal disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1)
HYPERNATREMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ILEUS (Gastrointestinal disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
SKIN INFECTION (Infections and infestations) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Carboplatin + Pemetrexed + Atezolizumab + Bevacizumab (N=30)
ABDOMINAL INFECTION (Infections and infestations) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8 (16)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (4)
ALLERGIC REACTION (Immune system disorders) | 2 (2)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 9 (10)
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 (1)
ANEMIA (Blood and lymphatic system disorders) | 18 (43)
ANOREXIA (Metabolism and nutrition disorders) | 12 (23)
ANOSMIA (Nervous system disorders) | 1 (1)
ANXIETY (Psychiatric disorders) | 5 (5)
AORTIC VALVE DISEASE (Cardiac disorders) | 1 (1)
ARTERIAL THROMBOEMBOLISM (Vascular disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 10 (11)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 9 (18)
ATRIAL FIBRILLATION (Cardiac disorders) | 5 (6)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 (16)
BELCHING (Gastrointestinal disorders) | 2 (2)
BLOATING (Gastrointestinal disorders) | 1 (1)
BLOOD AND LYMPHATIC SYSTEM DISORDERS (Blood and lymphatic system disorders) | 1 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 1 (1)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 2 (3)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1)
CARDIAC DISORDERS (Cardiac disorders) | 2 (2)
CARDIAC TROPONIN I INCREASED (Investigations) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1)
CHEST WALL PAIN (Musculoskeletal and connective tissue disorders) | 2 (3)
CHILLS (General disorders) | 1 (1)
CHOLESTEROL HIGH (Investigations) | 1 (1)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 2 (2)
COGNITIVE DISTURBANCE (Nervous system disorders) | 1 (1)
CONFUSION (Psychiatric disorders) | 2 (5)
CONJUNCTIVITIS INFECTIVE (Infections and infestations) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 21 (36)
COUGH (Respiratory, thoracic and mediastinal disorders) | 18 (21)
CREATININE INCREASED (Investigations) | 8 (14)
DEHYDRATION (Metabolism and nutrition disorders) | 7 (11)
DELIRIUM (Psychiatric disorders) | 1 (1)
DENTAL CARIES (Gastrointestinal disorders) | 2 (2)
DEPRESSION (Psychiatric disorders) | 8 (10)
DIARRHEA (Gastrointestinal disorders) | 12 (17)
DIZZINESS (Nervous system disorders) | 4 (4)
DRY EYE (Eye disorders) | 3 (3)
DRY MOUTH (Gastrointestinal disorders) | 1 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 (2)
DYSARTHRIA (Nervous system disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 8 (12)
DYSPEPSIA (Gastrointestinal disorders) | 5 (6)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 17 (21)
EAR PAIN (Ear and labyrinth disorders) | 1 (1)
EDEMA FACE (General disorders) | 3 (5)
EDEMA LIMBS (General disorders) | 11 (27)
EDEMA TRUNK (General disorders) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 6 (7)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 7 (11)
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 (2)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
EYE DISORDERS (Eye disorders) | 2 (4)
EYE PAIN (Eye disorders) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1)
FATIGUE (General disorders) | 27 (65)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
FEVER (General disorders) | 4 (5)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 3 (5)
FLATULENCE (Gastrointestinal disorders) | 2 (2)
FLUSHING (Vascular disorders) | 1 (2)
FOLLICULITIS (Infections and infestations) | 1 (2)
GASTRITIS (Gastrointestinal disorders) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 9 (10)
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 5 (5)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 5 (13)
GENERALIZED EDEMA (General disorders) | 2 (2)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 3 (3)
GINGIVAL PAIN (Gastrointestinal disorders) | 1 (1)
HALLUCINATIONS (Psychiatric disorders) | 1 (1)
HEADACHE (Nervous system disorders) | 10 (18)
HEARING IMPAIRED (Ear and labyrinth disorders) | 1 (1)
HEART FAILURE (Cardiac disorders) | 4 (4)
HEMATURIA (Renal and urinary disorders) | 1 (1)
HEMOGLOBINURIA (Renal and urinary disorders) | 2 (2)
HEMORRHOIDAL HEMORRHAGE (Gastrointestinal disorders) | 1 (2)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (3)
HERPES SIMPLEX REACTIVATION (Infections and infestations) | 1 (2)
HICCUPS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 3 (4)
HOT FLASHES (Vascular disorders) | 3 (3)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 9 (9)
HYPERKALEMIA (Metabolism and nutrition disorders) | 4 (4)
HYPERLIPIDEMIA (Metabolism and nutrition disorders) | 15 (15)
HYPERTENSION (Vascular disorders) | 24 (68)
HYPERTHYROIDISM (Endocrine disorders) | 6 (7)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 5 (13)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (16)
HYPOKALEMIA (Metabolism and nutrition disorders) | 5 (5)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 3 (6)
HYPONATREMIA (Metabolism and nutrition disorders) | 7 (8)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (5)
HYPOTENSION (Vascular disorders) | 1 (1)
HYPOTHYROIDISM (Endocrine disorders) | 7 (11)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
IMMUNE SYSTEM DISORDERS (Immune system disorders) | 1 (1)
INFECTIONS AND INFESTATIONS (Infections and infestations) | 1 (1)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (3)
INSOMNIA (Psychiatric disorders) | 16 (21)
INTRAOPERATIVE CARDIAC INJURY (Injury, poisoning and procedural complications) | 1 (1)
INVESTIGATIONS (Investigations) | 1 (1)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
LIPASE INCREASED (Investigations) | 3 (18)
LOCALIZED EDEMA (General disorders) | 3 (3)
LUNG INFECTION (Infections and infestations) | 3 (3)
LYMPHOCYTE COUNT DECREASED (Investigations) | 6 (6)
MANIA (Psychiatric disorders) | 1 (1)
METABOLISM AND NUTRITION DISORDERS (Metabolism and nutrition disorders) | 1 (1)
MITRAL VALVE DISEASE (Cardiac disorders) | 1 (1)
MOVEMENTS INVOLUNTARY (Nervous system disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 8 (21)
MUSCLE CRAMP (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER (Musculoskeletal and connective tissue disorders) | 5 (9)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 21 (74)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (2)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (4)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 1 (1)
NEURALGIA (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 9 (23)
NON-CARDIAC CHEST PAIN (General disorders) | 10 (13)
OPTIC NERVE DISORDER (Eye disorders) | 1 (1)
ORAL HEMORRHAGE (Gastrointestinal disorders) | 2 (3)
ORAL PAIN (Gastrointestinal disorders) | 1 (1)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 3 (3)
OTITIS EXTERNA (Infections and infestations) | 1 (1)
PAIN (General disorders) | 11 (34)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 8 (20)
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
PALPITATIONS (Cardiac disorders) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 1 (1)
PARESTHESIA (Nervous system disorders) | 1 (1)
PARONYCHIA (Infections and infestations) | 1 (1)
PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1)
PERIPHERAL ISCHEMIA (Vascular disorders) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 9 (18)
PHLEBITIS (Vascular disorders) | 4 (5)
PHLEBITIS INFECTIVE (Infections and infestations) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 6 (18)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 4 (5)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PROSTATIC OBSTRUCTION (Reproductive system and breast disorders) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 7 (19)
PRURITUS (Skin and subcutaneous tissue disorders) | 6 (11)
PSYCHIATRIC DISORDERS (Psychiatric disorders) | 1 (1)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 5 (10)
RECTAL HEMORRHAGE (Gastrointestinal disorders) | 1 (1)
RENAL AND URINARY DISORDERS (Renal and urinary disorders) | 1 (1)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS (Reproductive system and breast disorders) | 2 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS (Respiratory, thoracic and mediastinal disorders) | 5 (6)
RETINAL DETACHMENT (Eye disorders) | 1 (1)
RETINAL TEAR (Eye disorders) | 1 (1)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 2 (3)
SCALP PAIN (Skin and subcutaneous tissue disorders) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 6 (10)
SHINGLES (Infections and infestations) | 1 (3)
SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
SINUS TACHYCARDIA (Cardiac disorders) | 2 (2)
SINUSITIS (Infections and infestations) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 4 (6)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 2 (2)
SKIN INFECTION (Infections and infestations) | 1 (3)
SKIN ULCERATION (Skin and subcutaneous tissue disorders) | 1 (1)
SLEEP APNEA (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 1 (1)
STOMACH PAIN (Gastrointestinal disorders) | 2 (6)
SURGICAL AND MEDICAL PROCEDURES (Surgical and medical procedures) | 2 (2)
SYNCOPE (Nervous system disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 3 (3)
THRUSH (Infections and infestations) | 1 (1)
THYROID STIMULATING HORMONE INCREASED (Investigations) | 7 (9)
TINNITUS (Ear and labyrinth disorders) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 1 (2)
TREMOR (Nervous system disorders) | 1 (1)
TRICUSPID VALVE DISEASE (Cardiac disorders) | 1 (1)
TUMOR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4)
UPPER RESPIRATORY INFECTION (Infections and infestations) | 4 (4)
URINARY FREQUENCY (Renal and urinary disorders) | 3 (3)
URINARY RETENTION (Renal and urinary disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 5 (10)
VAGINAL DRYNESS (Reproductive system and breast disorders) | 1 (1)
VASCULAR DISORDERS (Vascular disorders) | 3 (4)
VENOUS INJURY (Injury, poisoning and procedural complications) | 1 (1)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1 (1)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 (2)
VERTIGO (Ear and labyrinth disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 13 (47)
WATERING EYES (Eye disorders) | 4 (6)
WEIGHT GAIN (Investigations) | 6 (10)
WEIGHT LOSS (Investigations) | 10 (16)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (3)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-07): https://cdn.clinicaltrials.gov/large-docs/44/NCT03713944/Prot_SAP_000.pdf